CLINICAL TRIAL: NCT06332118
Title: The Effect of Ice Massage Applied Before Arteriovenous Fistula Cannulation Procedure on Pain, Ecchymosis, Hematoma and Patient Satisfaction in Hemodialysis Patients
Brief Title: The Effect of Ice Massage on Pain, Ecchymosis, Hematoma and Patient Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Ercan Bakır, assoc prof, Erzurum Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: avf ice massage
Record Dates: First submitted 2024-03-04; First posted 2024-03-27 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; ice massage; pain; hematoma; ecchymosis; patient satisfaction
MeSH Terms: conditions — Pain; Hematoma; Ecchymosis; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The research is quasi-experimental and relationship-seeking in a pretest-posttest format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ice massage group (Experimental): Measurement surveys will be applied to obtain pre-test data from hemodialysis patients who meet the research criteria. After the preliminary test data are obtained, ice cubes prepared by the researchers before the needle insertion into the arteriovenous fistula for the hemodialysis procedure will be wrapped in a thin sponge and an ice massage will be applied to the needle insertion area of the patient in a direction that will not disrupt the circulation. This process will take approximately 3-5 minutes or the massage will be terminated when the patient feels drowsiness. In the next stage, the patient will undergo needle intervention for hemodialysis. At the end of this stage, the patient's pain will be evaluated. Patients will be re-evaluated at 24, 48 and 72 hours for ecchymosis and hematoma and relevant measurements will be provided.
  Interventions: Other: ice massage group

INTERVENTIONS:
Other: ice massage group — Measurement surveys will be applied to obtain pre-test data from hemodialysis patients who meet the research criteria. After the preliminary test data are obtained, ice cubes prepared by the researchers before the needle insertion into the arteriovenous fistula for the hemodialysis procedure will be wrapped in a thin sponge and an ice massage will be applied to the needle insertion area of the patient in a direction that will not disrupt the circulation. This process will take approximately 3-5 minutes or the massage will be terminated when the patient feels drowsiness. In the next stage, the patient will undergo needle intervention for hemodialysis. At the end of this stage, the patient's pain will be evaluated. Patients will be re-evaluated at 24, 48 and 72 hours for ecchymosis and hematoma and relevant measurements will be provided.

SUMMARY:
The research was planned to measure pain, ecchymosis, hematoma and patient satisfaction with ice massage applied to the fistula before the arteriovenous fistula procedure in hemodialysis patients. Patients who agree to participate in the study will be given ice massage before the procedure and the relevant parameters will be measured.

DETAILED DESCRIPTION:
Chronic renal failure is a condition that causes irreversible damage to kidney functions and prevents the excretion of metabolic wastes through urine. In the treatment of the disease; renal replacement therapies and kidney transplant options are available. The most commonly used treatment in end-stage renal failure patients is hemodialysis. Hemodialysis is performed through catheters and fistula channels. Patients receiving hemodialysis treatment through fistula are connected to the dialysis device. For this procedure, an injection occurs 2 or 3 times a week. It is a distressing situation for patients that needle insertion is painful during the procedure and that conditions such as ecchymosis and hematoma frequently occur afterwards. In this study, cold application was planned in a pre-test post-test design to evaluate pain, ecchymosis, hematoma and patient satisfaction. Volunteer participants who receive hemodialysis treatment through fistula will receive an ice massage for an average of 3-5 minutes on the fistula area where the needle will be inserted before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Conscious and oriented
* Communicable,
* Those who are 18 years or older,
* Hemodialysis treatment is applied via arteriovenous fistula,
* There are no signs of infection such as redness, swelling, or open wound in the area where the procedure will be performed,
* Patient: International Normalized Ratio: 2-3, Activated Partial Thromboplastin Time: 27-45 sec. Prothrombin Time: 11-16 sec. Thrombocyte: 125-350 m3
* Can tolerate the application,
* 10 minutes before starting Hemodialysis treatment. vissual analog scale pain score was evaluated beforehand and vissual analog scale was ≥4.
* Patients who agree to participate in the study verbally and in writing will be included in the research.

Exclusion Criteria:

* Unconscious,
* Unable to communicate,
* Those who are under 18 years of age,
* Hemodialysis treatment is not applied via arteriovenous fistula,
* If there is any sign of infection such as redness, swelling, open wound in the area where cannulation will be performed,
* 10 minutes before starting hemodialysis treatment. vissual analog scale pain score was evaluated beforehand and vissual analog scale ≤ 4
* Using any painkillers before the procedure on the same day,
* Patient: International Normalized Ratio: 2-3, Activated Partial Thromboplastin Time: 27-45 sec. Prothrombin Time: 11-16 sec. Thrombocyte: above 125-350 m3, prone to bleeding,
* Patients who cannot tolerate the application or do not want to participate in the study voluntarily will not be included in the research.

Exclusion Criteria:

Patients who cannot tolerate ice massage during the procedure will not be included in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 3 days
  Vissual analog scale: The scale is rated between 0 points and 10 points. 0 indicates that the patient has no pain, and 10 indicates that the patient has unbearable pain. Patients report their pain status on a scale of 0 to 10 points.

SECONDARY OUTCOMES:
Ecchymosis degree | 3 days
  The area of the ecchymosis will be calculated in square millimeters with polyethylene millimetric plastic film (opsite flexigrid).
Hematoma degree | 3 days
  The area of the hematoma will be calculated in square millimeters with polyethylene millimetric plastic film (opsite flexigrid).
Patient satisfaction score | 3 days
  Numerical Satisfaction Scale: The scale is rated between 0 points and 10 points. 0 indicates that the patient is very dissatisfied, and 10 indicates that the patient is very satisfied. Patients report their satisfaction between 0 and 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bakır, PhD, Study Director — erzurum tecnical university
Locations (1):
- Ercan Bakır, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koushki B, Khajeh M, Bagheri H, Talebi SS, Ebrahimi H. Comparing the Effect of Local Application of Peppermint and Cold Compresses on the Severity of Pain from Venipuncture in Dialysis Patients: A Parallel Randomized Clinical Trial Study. Saudi J Kidney Dis Transpl. 2023 Jul 1;34(4):288-296. doi: 10.4103/1319-2442.395444. Epub 2024 Feb 12. PMID 38345583
- [Background] Ghoreyshi Z, Amerian M, Amanpour F, Ebrahimi H. Evaluation and comparison of the effects of Xyla-P cream and cold compress on the pain caused by the cannulation of arteriovenous fistula in hemodialysis patients. Saudi J Kidney Dis Transpl. 2018 Mar-Apr;29(2):369-375. doi: 10.4103/1319-2442.229265. PMID 29657205
- [Background] Kesik G, Ozdemir L, Yildirim T, Jabrayilov J, Celiksoz G. Effects of warm or cold compresses applied to the legs during hemodialysis on cramps, fatigue, and patient comfort: A placebo-controlled randomized trial. Hemodial Int. 2023 Apr;27(2):117-125. doi: 10.1111/hdi.13070. Epub 2023 Feb 14. PMID 36788410
- [Background] Dehghan M, Hosseini SJ, Shahrbabaki PM, Forouzi MA, Roy C. The Effect of Acupressure and Cryotherapy on the Pain of Patients on Hemodialysis During Arteriovenous Fistula Cannulation: A Randomized Crossover Clinical Trial. Nephrol Nurs J. 2023 Mar-Apr;50(2):131-139. PMID 37074938
- [Background] Al Amer HS, Dator WL, Abunab HY, Mari M. Cryotherapy intervention in relieving arteriovenous fistula cannulation-related pain among hemodialysis patients at the King Khalid Hospital, Tabuk, Kingdom of Saudi Arabia. Saudi J Kidney Dis Transpl. 2017 Sep-Oct;28(5):1050-1056. doi: 10.4103/1319-2442.215141. PMID 28937062